CLINICAL TRIAL: NCT05050071
Title: Comparative Evaluation of Antibacterial Effect of Allium Sativum, Calcium Hydroxide and Their Combination as Intracanal Medicaments in Infected Mature Teeth. A Randomized Control Trial
Brief Title: Evaluation of Antibacterial Effect of Allium Sativum, Calcium Hydroxide and Their Combination in Infected Mature Teeth
Acronym: Garlic
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Reham Mohamed, Principle Investigator, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 228/2019
Record Dates: First submitted 2021-08-12; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Drug Effect
Keywords: Calcium hydroxide; Enterococcus faecalis; Garlic; Intra-canal medication; Streptococcus; Quantitative real-time polymerase chain reaction
MeSH Terms: interventions — Calcium Hydroxide; Polymerase Chain Reaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (6):
- Calcium hydroxide (7 days) (Active Comparator): is also known as slaked lime or calcium hydrate. It is produced by the hydration of lime
  Interventions: Drug: Allium Sativum; Device: Polymerase chain reaction
- Allium sativum (7 days) (Experimental): is a species of bulbous flowering plant in the onion genus Allium
  Interventions: Drug: Allium Sativum; Device: Polymerase chain reaction
- Combination (7 days) (Experimental): combination between Calcium hydroxide and Allium sativum
  Interventions: Drug: Allium Sativum; Device: Polymerase chain reaction
- Calcium hydroxide (14 days) (Active Comparator): is also known as slaked lime or calcium hydrate. It is produced by the hydration of lime
  Interventions: Drug: Allium Sativum; Device: Polymerase chain reaction
- Allium sativum (14 days) (Experimental): is a species of bulbous flowering plant in the onion genus Allium
  Interventions: Drug: Allium Sativum; Device: Polymerase chain reaction
- Combination (14 days) (Experimental): combination between Calcium hydroxide and Allium sativum
  Interventions: Drug: Allium Sativum; Device: Polymerase chain reaction

INTERVENTIONS:
Drug: Allium Sativum — Sixty-six permanent mature necrotic incisors associated with apical periodontitis in male children were selected. Teeth were randomly divided into three groups (n=22) according to intra canal medications used; group I: Ca OH2, group II: garlic extract and group III: mixture of Ca OH2 and garlic extract. After access preparation, four microbiological samples (S) were as follows; (S1): were taken before canal instrumentation and irrigation. (S2): after cleaning and shaping, Then, the third samples (S3) and forth samples (S4) were taken after placement of the tested intracanal medications into the corresponding canals, for 7 and 14 days respectively. Total DNA was extracted from microbiological samples and relative quantitive real time PCR reactions were done to quantify the relative gene expression levels (FC) for Streptococcus and Enterococcus faecalis species.
  Other Names: Combination of Allium Sativum and Calcium hydroxide; Calcium hydroxide
Device: Polymerase chain reaction — Change in the bacterial load in response to different treatment procedures

SUMMARY:
This study was to evaluate and compare garlic extract antibacterial effect when used as an intra-canal medicament in infected mature anterior teeth with calcium hydroxide and a mixture of calcium hydroxide and garlic, using real time PCR analysis.

DETAILED DESCRIPTION:
Sixty-six permanent mature necrotic incisors associated with apical periodontitis in male children were selected. Teeth were randomly divided into three groups (n=22) according to intra canal medications used; group I: Ca OH2, group II: garlic extract and group III: mixture of Ca OH2 and garlic extract. After access preparation, four microbiological samples (S) were taken using sterile absorbent paper points as follows; (S1): were taken before canal instrumentation and irrigation. (S2): after cleaning and shaping, Then, the third samples (S3) and forth samples (S4) were taken after placement of the tested intracanal medications into the corresponding canals, for 7 and 14 days respectively. Total DNA was extracted from microbiological samples and relative quantitive real time PCR reactions were done to quantify the relative gene expression levels (FC) for Streptococcus and Enterococcus faecalis species. Data was statistically analyzed using Kruskal-Wallis and Freidman's tests, followed by Mann-Whitney and Wilcoxon singed rank tests at significance level p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Cooperative male children with age ranging from 10 to 13 years.
2. All patients should have pulp necrosis with apical periodontitis in one or more upper incisor(s).
3. Teeth included in the study were preliminarily evaluated by preoperative periapical radiographs and should have: single canal (type I vertucci's classification) with closed apices, periapical lesions of endodontic origin with a diameter ranging from 2 to 5 mm without any previous RCT procedure.

Exclusion Criteria:

1. immune-compromised patient or patient with complicating systemic disease.
2. Patients received antibiotic therapy within the previous 3 months.
3. Tooth having gross carious lesions, fractures or cracks involving the periodontium (un-restorable tooth).
4. Tooth with root canal calcifications or resorption

6- Tooth with periodontal pockets of more than 4 mm depth, with or without endo-perio communication either concomitant or combined.

Ages: 10 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Test the antibacterial efficiency of Garlic extract as intracanal medicament in comparison to Calcium hydroxide and their combinations , against E.faecalis and streptococcus bacteria using qRT-PCR analysis. | 12 months
  The change in the mean relative gene expression (bacterial load), for E.faecalis and streptococcus species was measured using quantitative real time polymerase chain reaction (qRT-PCR) after placement garlic (Allium Sativum), Calcium hydroxide and their combinations for one week, in infected single rooted anterior teeth. Statistical analysis was done to compare between the tested medicaments

SECONDARY OUTCOMES:
Test the antibacterial effect of increasing the contact time (14 days) for garlic (Allium Sativum), Calcium hydroxide or their combinations inside infected root canals, against E.faecalis and streptococcus bacteria using qRT-PCR analysis. | 12 months
  The change in the mean relative gene expression (bacterial load), for E.faecalis and streptococcus species was measured using quantitative real time polymerase chain reaction (qRT-PCR) after placement garlic (Allium Sativum), Calcium hydroxide and their combinations for two weeks, in infected single rooted anterior teeth. Statistical analysis was done to compare between the tested medicaments.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa M. Mahfouz, PhD, Principal Investigator — Suez Canal University, Ismailia, Egypt
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Protocol & Conclusion
Supporting Information: Study Protocol, SAP
Time Frame: for 1 month
URL: http://suez.edu.eg